CLINICAL TRIAL: NCT04003337
Title: Selection of the Embryo to Transfer by Morphokinetics vs. Morphological Evaluation. Prospective and Randomized Trial of Patients Using Time-lapse (Embryoscope®).
Brief Title: Selection of the Embryo to Transfer by Morphokinetics vs. Morphological Evaluation.
Acronym: EmbryoSEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Procreatec (Other)
Collaborators: Sociedad Espanola Fertilidad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EmbryoSEL
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Embryo Implantation
MeSH Terms: interventions — Fetoscopes

STUDY DESIGN:
Intervention Model Description: Two arms interventional prospective randomized controlled trial.
Who Masked: Participant, Care Provider
Masking Description: Once patients accept to be enrolled in the study, one of the nurses will allocate the patient to one of study groups. Neither the patient nor the doctor will know the group assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A: Morphological embryo selection (No Intervention): Patients enrolled in group A will receive an embryo transfer according to classical morphological criteria.
- GROUP B: Morpho-kinetics embryo selection (Active Comparator): Patients enrolled in group B will receive an embryo transfer according to new morphokinetics criteria.
  Interventions: Other: Morpho-kinetics selection with time-lapse (Embryoscope) evaluation

INTERVENTIONS:
Other: Morpho-kinetics selection with time-lapse (Embryoscope) evaluation — Embryos in group B will be selected in blastocyst stage according to morpho-kinetics criteria before the embryo transfer
  Arms: GROUP B: Morpho-kinetics embryo selection

SUMMARY:
Our study intends to demonstrate that the selection of an embryo to transfer it at the sage of blastocyst through morphokinetics (analysis of embryos depending not only in their morphology -that is, the aspect of the embryo-, but also based on times of cell division) during the use of time-lapse (Embryoscope®) may have a better impact in clinical results, as selection is not performed in mere morphological evolution (visual aspect of the embryo) of the embryos.

DETAILED DESCRIPTION:
Our study intends to demonstrate that the selection of an embryo to transfer it at the sage of blastocyst through morphokinetics (analysis of embryos depending not only in their morphology -that is, the aspect of the embryo-, but also based on times of cell division) during the use of time-lapse (Embryoscope®) may have a better impact in clinical results, as selection is not performed in mere morphological evolution (visual aspect of the embryo) of the embryos.

In order to obtain this objective, patients participating in the study will be randomly assigned to one of the following groups:

Group A: Patients who will perform an embryo transfer of a blastocyst using morphological criteria to evaluate que quality of the blastocyst (Gardner Classification), that is, based on the aspect or form of the embryo.

Group B: Patients who will perform an embryo transfer of a blastocyst using morphokinetics criteria to evaluate the quality of the blastocyst (Embryoscope®), that is, based not only in the aspect of the embryo but also in cell division times experimented by the embryos.

ELIGIBILITY:
Inclusion Criteria:

* Egg-donation IVF patients
* IVF patients if < 38 years
* Sperm concentration > 2 million/ml
* Frozen eggs for
* Single embryo transfer
* ICSI fertilization

Exclusion Criteria:

* Uterine pathologies that may interfere with implantation
* Endometriosis
* Frozen eggs
* Pre implantation genetic testing of the embryos
* Day 3 embryo transfer
* Conventional IVF treatments

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Estimated)
Dates: Start 2017-01-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Rate | 12-14 days after the embryo transfer
  Positive pregnancy test

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | 12-15 days after the positive blood test for pregnancy
  US pregnancy confirmation

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Lopez, Principal Investigator — Procreatec
Locations (1):
- Procreatec, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided